CLINICAL TRIAL: NCT01270958
Title: A Phase-IV, Open-label Study to Evaluate Safety/Tolerability of Once-daily AVAMYS (TM) Aqueous Nasal Spray 110mcg Among Vietnamese Adult Patients With Established Perennial Allergic Rhinitis (PAR)
Brief Title: A Phase-IV, Open-label Study to Evaluate Safety/Tolerability of Once-daily AVAMYS (TM) Aqueous Nasal Spray 110mcg Among Vietnamese Adult Patients With Established Perennial Allergic Rhinitis
Acronym: AVY-REG00108VN
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 112185
Record Dates: First submitted 2010-08-31; First posted 2011-01-05 (Estimated); Results first posted 2011-01-05 (Estimated); Last update posted 2014-08-06 (Estimated); Status verified 2014-08

CONDITIONS: Rhinitis, Allergic, Perennial
Keywords: AVY-REG00108VN
MeSH Terms: conditions — Rhinitis, Allergic, Perennial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TREATMENT (Experimental): 50 adult patients with Perennial Allergic Rhinities treated with Avamys.
  Interventions: Drug: Avamys aqueous nasal spray 110mcg

INTERVENTIONS:
Drug: Avamys aqueous nasal spray 110mcg — At the visit 1, subjects who fulfill the inclusion criteria are eligible to be included in the group to self-administer intranasal treatment of fluticasone furoate aqueous nasal spray 110 mcg once daily for 6 week. The subjects are instructed to administer two sprays from the device into each nostril once daily every morning. Administration of the dose will be performed by alternately spraying one spray to each nostril followed by a second spray to each nostril. Subjects will not be permitted to take any anti-allergy or rhinitis medication during the screening or treatment period.
  Throughout the study, subjects will document their study drug administration/compliance, any medical conditions experienced, and any concomitant medications taken.

SUMMARY:
Allergic rhinitis is an IgE-mediated, inflammatory disorder of the upper airway that occurs following allergen exposure. Perennial Allergic Rhinitis (PAR) starts in early childhood and occurs all year around. It's caused by allergy to the aerosolised droppings of house dust mites and pet skin flakes (dander). Occasionally, indoor mould spores and, in rare cases, food allergy can be causes.

Intranasal corticosteroids are highly effective medications for controlling the nasal symptoms that accompany allergic rhinitis.

AVAMYS (TM) (fluticasone furoate aqueous nasal spray 100mcg) has been shown having effects on nasal symptoms of seasonal and perennial allergic rhinitis and on the ocular symptoms of allergic rhinitis and has been evaluated as effective and safe for treatment seasonal and perennial allergic rhinitis by FDA. It is speculated that AVAMYS (TM) is also effective and safe for Vietnamese patients. However before being used widely for patients across the country, AVAMYS (TM) should be proved that it is safe for Vietnamese patients.

The objective of this study is to evaluate the safety of fluticasone furoate aqueous nasal spray 110mcg once daily in adults with PAR.

This is a 6-week, open trial. A study center will be enlisted to recruit a minimum of 50 PAR subjects.

At the visit 1, subjects who fulfill the inclusion criteria are eligible to be included in the group to self-administer intranasal treatment of fluticasone furoate aqueous nasal spray 110 mcg once daily for 6 week. The subjects are instructed to administer two sprays from the device into each nostril once daily every morning. Administration of the dose will be performed by alternately spraying one spray to each nostril followed by a second spray to each nostril. Subjects will not be permitted to take any anti-allergy or rhinitis medication during the screening or treatment period.

Throughout the study, subjects will document their study drug administration/compliance, any medical conditions experienced, and any concomitant medications taken. All subjects are outpatients.

The safety assessments include a summary of the frequency and type of clinical adverse events that occur during the study. In addition, hematology and chemistry analyses of blood samples are also implemented. A physical examination and nasal examination are also performed and vital signs collected. Twelve-lead ECGs are performed at all visits.

DETAILED DESCRIPTION:
Rationale Allergic rhinitis is an IgE-mediated, inflammatory disorder of the upper airway that occurs following allergen exposure. Perennial Allergic Rhinitis (PAR) starts in early childhood and occurs all year around. It's caused by allergy to the aerosolised droppings of house dust mites and pet skin flakes (dander). Occasionally, indoor mould spores and, in rare cases, food allergy can be causes.

Intranasal corticosteroids are highly effective medications for controlling the nasal symptoms that accompany allergic rhinitis.

AVAMYS (TM) (fluticasone furoate aqueous nasal spray 100mcg) has been shown having effects on nasal symptoms of seasonal and perennial allergic rhinitis and on the ocular symptoms of allergic rhinitis and has been evaluated as effective and safe for treatment seasonal and perennial allergic rhinitis by FDA. It is speculated that AVAMYS (TM) is also effective and safe for Vietnamese patients. However before being used widely for patients across the country, AVAMYS (TM) should be proved that it is safe for Vietnamese patients.

Objective(s) The objective of this study is to evaluate the safety of fluticasone furoate aqueous nasal spray 110mcg once daily in adults with PAR.

As treatment duration of duration of PAR is normally longer than that of SAR, the safety/tolerability evaluation of PAR treatment is well sufficient for the similar evaluation of SAR.

Safety Endpoints

* Frequency of solicited clinical adverse events (headache, epistaxis, pharyngolaryngeal pain)
* Vital signs (systolic and diastolic blood pressure, heart rate [pulse])
* Clinical laboratory tests at baseline, during and at study termination, specifically as follows:

Chemistry: Glucose, ALT & AST, Total Bilirubin, Alkaline phosphatase, Total Protein & Albumin Hematology: Complete Blood Count (CBC) Pregnancy test: Urine pregnancy test for all female subjects at Screening, Visit 2 & Visit 3.

• 12-lead electrocardiograms (ECGs) at baseline and at study termination

Study Design This is a 6-week, open trial. A study center will be enlisted to recruite a minimum of 50 PAR subjects. At the visit 1, subjects who fulfil the inclusion criteria are eligible to be include in the group to self-administer intranasal treatment of fluticasone furoate aqueous nasal spray 110 mcg once daily for 6 week. The subjects are instructed to administer two sprays from the device into each nostril once daily every morning. Administration of the dose will be performed by alternately spraying one spray to each nostril followed by a second spray to each nostril. Subjects will not be permitted to take any anti-allergy or rhinitis medication during the screening or treatment period.

Throughout the study, subjects will document their study drug administration/compliance, any medical conditions experienced, and any concomitant medications taken. All subjects are outpatients. Clinic visits for a study subject are scheduled to occur at the following intervals:

Screening visit: To collect Inform Consent Form and evaluate eligibility, medical history, clinical status, electrocardiography and necessary laboratory testing. If a subject is eligible and is not on any anti-histamin medications, he/she can enter the study right at this visit (i.e. on study medication).

Visit 1: Three to five days after the screening visit. This visit is due to a subject who is eligible and is on an anti-histamin medication at the screening visit. The subject must have been discontinued the anti-histamin medication(s) since the screening visit. He/she is then clinically evaluated, prescribed with study drug and instructed how to fill the Diary Card.

Visit 2: Fourteen ( ± 1) day after Visit 1 or Day 15. Clinical evaluation, drug accountability, Diary card collection and study-specific laboratory testings are applied.

Visit 3: Forty-two ( ± 1) day after Visit 1. Clinical evaluation, drug accountability, Diary card collection and study-specific laboratory testings are applied. All study information in the Case Report Form (CRF) of the subject is reviewed. A PAR subject is considered to fulfill the study only when this visit is completed.

A follow-up telephone contact is made 3 to 5 days after Visit 3/Early Withdrawal to assess for any adverse effects after discontinuing study treatment.

Study Population A minimum of 50 adults with perennial allergic rhinitis (PAR) are recruited for this study.

Study Assessments The safety assessments include a summary of the frequency and type of clinical adverse events that occur during the study. In addition, hematology and chemistry analyses of blood samples are also implemented. A physical examination and nasal examination are also performed and vital signs collected. Twelve-lead ECGs are performed at all visits.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent: Subject has provided an appropriately signed and dated informed consent.
2. Outpatient: Subject is treatable on an outpatient basis.
3. Age ≥ 18 years at Visit 1
4. Male or eligible female: To be eligible for entry into the study, females of childbearing potential must commit to the consistent and correct use of an acceptable method of birth control, as defined by the following:

   * Male partner who is sterile prior to the female subject's entry into the study and is the sole sexual partner for that female subject
   * Implants of levonorgestrel
   * Injectable progestogen
   * Oral contraceptive (either combined estrogen/progestin or progestin only)
   * Any intrauterine device (IUD) with a documented failure rate of less than 1% per year, or
   * Double barrier method - spermacide plus a mechanical barrier (e.g., spermacide plus a male condom or a spermacide and female diaphragm).

   Females of childbearing potential who are not sexually active must commit to complete abstinence from intercourse for two weeks before exposure to the study drug, throughout the clinical trial, and for a period after the trial to account for elimination of the drug (minimum of six days).

   Female subjects should not be enrolled if they plan to become pregnant during the time of study participation. A urine pregnancy test is performed at the screening visit and the final visit.
5. Diagnosis of perennial allergic rhinitis (PAR)

   * Documented clinical history of PAR, if available, with perennial allergy symptoms during each of the last two years
   * A positive skin test (by prick method) to testing allergens within 12 months prior to or at screening visit.

   A positive skin test is defined as a wheal ≥3 mm larger than the diluent control for prick testing.

   Subjects who meet the above criteria and who may also have perennial allergic rhinitis or vasomotor rhinitis are eligible for entry to the study.
6. Ability to comply with study procedures: Subject understands and is willing, able and likely to comply with study procedures and restrictions.
7. Literate: Subject must be able to read, comprehend, and record information in Vietnamese.

Exclusion Criteria:

A subject is not eligible for inclusion in this study if any of the following criteria applies.

1. Significant concomitant medical condition(s), defined as but not limited to:

   1. Historical or current evidence of a clinically significant uncontrolled disease of any body system (e.g., tuberculosis, psychological disorders, eczema). Significant is defined as any disease that, in the opinion of the investigator, would put the safety of the subject at risk through study participation or which would confound the interpretation of the study results if the disease/condition exacerbated during the study.
   2. A severe physical obstruction of the nose (e.g., deviated septum or nasal polyp) or nasal septal perforation that could affect the deposition of intranasal study drug.
   3. Nasal (eg, nasal septum), ocular, or throat injury or surgery in the last 3 months
   4. Asthma at all severities
   5. Rhinitis medicamentosa
   6. Bacterial or viral infection (e.g., common cold) of the eyes or upper respiratory tract within two weeks of Screening visit or during the screening period
   7. Documented evidence of acute or significant chronic sinusitis, as determined by the individual investigator.
   8. Current or history of glaucoma and/or cataracts or ocular herpes simplex
   9. Physical impairment that would affect subject's ability to participate safely and fully in the study
   10. Clinical evidence of a Candida infection of the nose
   11. History of psychiatric disease, intellectual deficiency, poor motivation, substance abuse (including drug and alcohol) or other conditions that will limit the validity of informed consent or that would confound the interpretation of the study results
   12. History of adrenal insufficiency
2. Use of corticosteroids, defined as:

   * Intranasal corticosteroid within four weeks prior to Screening visit or Visit 1.
   * Inhaled, oral, intramuscular, intravenous, ocular, and/or dermatological corticosteroid (with the exception of hydrocortisone cream/ointment, 1% or less) within eight weeks prior to Screening visit or Visit 1.
3. Use of other allergy medications within the timeframe indicated relative to Screening visit or Visit 1

   * Intranasal or ocular cromolyn within 2 weeks prior to Screening visit or Visit 1
   * Long-acting antihistamines within 10 days prior to Screening visit or Visit 1 (e.g., loratadine, desloratadine, fexofenadine, cetirizine)
   * Intranasal antihistamines (e.g. Astelin‡ ) within 2 weeks prior to Screening visit or Visit 1
   * Oral or intranasal decongestants within three days prior to Screening visit or Visit 1
4. Use of any medications that significantly inhibit the cytochrome P450 subfamily enzyme CYP3A4, including ritonavir and ketoconazole.
5. Contact Lens and Ocular Preparations: Subjects are not permitted to wear contact lens or use any ocular preparations, including artificial tears, eyewash/ irrigation solutions, or lubricants, during the screening and treatment periods. No exclusion period prior to screening (Visit 1) is required for these ocular products. Eye glasses are permitted during the study.
6. Allergy/Intolerance: Known hypersensitivity to corticosteroids or any excipients in the product
7. Clinical trial/experimental medication experience

   * Has recent exposure to an investigational study drug within 30 days of Visit 1
   * Participation in a previous study of intranasal fluticasone furoate
8. Positive pregnancy test or female who is breastfeeding: Has a positive or inconclusive pregnancy test at Screening visit or Visit 1
9. Affiliation with investigational site: Subject is a participating investigator, sub-investigator, study co-ordinator, or employee of a participating investigator, or is an immediate family member of the aforementioned.
10. Current tobacco use: Subjects who have used smoking products including cigarettes, cigars, and pipe or chewing tobacco within the past year.
11. Findings of a clinically significant, abnormal ECG.
12. Findings of a clinically significant laboratory abnormality.
13. Chickenpox or measles: A subject is not eligible if he/she currently has chickenpox or measles, or has been exposed to chickenpox or measles during the last three weeks and is nonimmune. If a subject develops chickenpox or measles during the study, he/she will be withdrawn from the study. If a non-immune subject is exposed to chickenpox or measles during the study, his/her continuation in the study will be at the discretion of the investigator, taking into consideration the likelihood of developing active disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-08; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Hà Nội, Vietnam

REFERENCES:
- [Background] Vo Thanh Quang, Pham Tuan Canh, Nguyen Nhat Linh. A phase IV, open-label study to evaluate safety/tolerability of once-daily AVAMYSTM aqueous nasal spray 110 mcg among Vietnamese adult patients with established perennial allergic rhinitis (PAR). 2011;2(2):56-4.

RESULTS

PARTICIPANT FLOW:
Groups:
- Fluticasone Furoate 110 mcg: Fluticasone furoate 110 micrograms (mcg) self-administered intranasally once daily
Period: Overall Study
Arm/Group | Fluticasone Furoate 110 mcg
Started | 60
Completed | 56
Not Completed | 4
Not completed — Lost to Follow-up | 2
Not completed — Did not meet inclusion criteria for age | 2

BASELINE CHARACTERISTICS:
Arm/Group | Fluticasone Furoate 110 mcg
Number analyzed (Participants) | 60
Age, Continuous [Mean (Standard Deviation); unit: Years] | 35.5 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 27
Race/Ethnicity, Customized [Number; unit: participants]
  Vietnamese | 60
  Other | 0

OUTCOME MEASURES:

1. Primary Outcome: Systolic Blood Pressure at Screening/Visit 1, Visit 2, and Visit 3
Description: Blood pressure (BP) is the pressure exerted by circulating blood upon the walls of blood vessels. During each heartbeat, BP varies between a maximum (systolic) and a minimum (diastolic) pressure.
Time Frame: Screening/Visit 1 (3-5 days after Screening Visit), Visit 2 (14 [± 1] days after Visit 1, or Day 15), and Visit 3 (42 [± 1] days after Visit 1, or Day 43)
Population: Intent-to-Treat (ITT) Population: all participants who received at least one dose of study drug. Some participants were lost to follow-up and may not have been dosed with study drug.
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | Fluticasone Furoate 110 mcg
Number analyzed (Participants) | 56
millimeters of mercury (mmHg)
  Screening/Visit 1 | 110.98 (9.23)
  Visit 2 | 110.63 (11.69)
  Visit 3 | 110.00 (11.61)
Statistical Analysis 1: Comparison: Fluticasone Furoate 110 mcg; Test type: Superiority or Other; p > 0.05, t-test, 2 sided — Comparison between Screening value and Visit 3 value

2. Primary Outcome: Diastolic Blood Pressure at Screening/Visit 1, Visit 2, and Visit 3
Description: as for outcome 1
Time Frame: as for outcome 1
Population: ITT Population: Some participants were lost to follow-up and may not have been dosed with study drug.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Fluticasone Furoate 110 mcg
Number analyzed (Participants) | 56
mmHg
  Screening/Visit 1 | 70.36 (6.6)
  Visit 2 | 71.79 (6.37)
  Visit 3 | 70.63 (6.69)
Statistical Analysis 1: Comparison: Fluticasone Furoate 110 mcg; Test type: Superiority or Other; p > 0.05, t-test, 2 sided — Comparison between Screening value and Visit 3 value

3. Primary Outcome: Heart Rate at Screening/Visit 1, Visit 2, and Visit 3
Description: Heart rate is measured as the number of heart beats per unit time.
Time Frame: as for outcome 1
Population: ITT Population
Measure: Mean (Standard Deviation); unit: beats per minute (bpm)
Arm/Group | Fluticasone Furoate 110 mcg
Number analyzed (Participants) | 56
beats per minute (bpm)
  Screening/Visit 1 | 72.80 (7.70)
  Visit 2 | 73.95 (6.39)
  Visit 3 | 73.04 (6.61)
Statistical Analysis 1: Comparison: Fluticasone Furoate 110 mcg; Test type: Superiority or Other; p > 0.05, t-test, 2 sided — Comparison between Screening value and Visit 3 value

4. Primary Outcome: Hemoglobin Values at Baseline and After Treatment Completion
Description: Hemoglobin functions primarily to transport oxygen from the lungs to the body tissues. Normal range: 125-160 grams per liter (g/L).
Time Frame: Baseline and treatment completion (up to Week 6)
Population: ITT Population
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Fluticasone Furoate 110 mcg
Number analyzed (Participants) | 56
g/L
  Baseline | 137.20 (12.06)
  After treatment completion | 136.16 (10.82)
Statistical Analysis 1: Comparison: Fluticasone Furoate 110 mcg; Test type: Superiority or Other; p > 0.05, t-test, 2 sided — Comparison between Screening value and Visit 3 value

5. Primary Outcome: Hematocrit Values at Baseline and After Treatment Completion
Description: Hematocrit is the proportion of blood volume that is occupied by red blood cells. The hematocrit (Hct) is expressed as liter of red blood cells in liters of blood. Normal range: 0.35-0.50 Liter/Liter.
Time Frame: Baseline and treatment completion (up to Week 6)
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Liter/Liter
Arm/Group | Fluticasone Furoate 110 mcg
Number analyzed (Participants) | 56
Liter/Liter
  Baseline | 0.40 (0.03)
  After treatment completion | 0.40 (0.03)
Statistical Analysis 1: Comparison: Fluticasone Furoate 110 mcg; Test type: Superiority or Other; p > 0.05, t-test, 2 sided — Comparison between Screening value and Visit 3 value

6. Primary Outcome: Red Blood Cell Count at Baseline and After Treatment Completion
Description: Red blood cells are cells in the blood that are used to transport oxygen throughout the body. Normal range: 3.9-5.8 10^12 cells per liter (Tetra/L).
Time Frame: Baseline and treatment completion (up to Week 6)
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Tetra/L
Arm/Group | Fluticasone Furoate 110 mcg
Number analyzed (Participants) | 56
Tetra/L
  Baseline | 4.49 (0.40)
  After treatment completion | 4.45 (0.36)
Statistical Analysis 1: Comparison: Fluticasone Furoate 110 mcg; Test type: Superiority or Other; p > 0.05, t-test, 2 sided — Comparison between Screening value and Visit 3 value

7. Primary Outcome: White Blood Cell Count at Baseline and After Treatment Completion
Description: White blood cells are cells of the immune system that defend the body against both infectious disease and foreign materials. Normal range: 4-10 10^9 cells per liter (Giga/L).
Time Frame: Baseline and treatment completion (up to Week 6)
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Giga/L
Arm/Group | Fluticasone Furoate 110 mcg
Number analyzed (Participants) | 56
Giga/L
  Baseline | 7.29 (1.76)
  After treatment completion | 7.08 (1.32)
Statistical Analysis 1: Comparison: Fluticasone Furoate 110 mcg; Test type: Superiority or Other; p > 0.05, t-test, 2 sided — Comparison between Screening value and Visit 3 value

8. Primary Outcome: Platelet Count at Baseline and After Treatment Completion
Description: Platelets are cells found in the blood that play a role in blood clotting. Normal range: 150-400 Giga/L.
Time Frame: Baseline and treatment completion (up to Week 6)
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Giga/L
Arm/Group | Fluticasone Furoate 110 mcg
Number analyzed (Participants) | 56
Giga/L
  Baseline | 259.80 (59.02)
  After treatment completion | 255.16 (49.57)
Statistical Analysis 1: Comparison: Fluticasone Furoate 110 mcg; Test type: Superiority or Other; p > 0.05, t-test, 2 sided — Comparison between Screening value and Visit 3 value

9. Primary Outcome: Sodium Count at Baseline and After Treatment Completion
Description: Sodium is the major positive ion (cation) found outside of cells. The balance of the electrolytes in our bodies is essential for normal function of our cells and our organs. Normal range: 135-145 millimoles per liter (mmol/L).
Time Frame: Baseline and treatment completion (up to Week 6)
Population: ITT Population
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Fluticasone Furoate 110 mcg
Number analyzed (Participants) | 56
mmol/L
  Baseline | 138.09 (1.58)
  After treatment completion | 139.13 (1.95)
Statistical Analysis 1: Comparison: Fluticasone Furoate 110 mcg; Test type: Superiority or Other; p < 0.01, t-test, 2 sided — Comparison between Screening value and Visit 3 value

10. Primary Outcome: Potassium Count at Baseline and After Treatment Completion
Description: Potassium is the major positive ion (cation) found inside of cells. The balance of the electrolytes in our bodies is essential for normal function of our cells and our organs. Normal range: 3.5-5.0 mmol/L.
Time Frame: Baseline and treatment completion (up to Week 6)
Population: ITT Population
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Fluticasone Furoate 110 mcg
Number analyzed (Participants) | 56
mmol/L
  Baseline | 3.84 (0.27)
  After treatment completion | 3.90 (0.02)
Statistical Analysis 1: Comparison: Fluticasone Furoate 110 mcg; Test type: Superiority or Other; p > 0.05, t-test, 2 sided — Comparison between Screening value and Visit 3 value

11. Primary Outcome: Total Bilirubin Value at Baseline and After Treatment Completion
Description: Total bilirubin is formed when hemoglobin breaks down. Bilirubin is excreted in bile and urine, and elevated levels may indicate certain diseases. Normal range: <=17 micromoles per liter (umol/L).
Time Frame: Baseline and treatment completion (up to Week 6)
Population: ITT Population
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Fluticasone Furoate 110 mcg
Number analyzed (Participants) | 56
umol/L
  Baseline | 11.91 (3.74)
  After treatment completion | 13.54 (12.39)
Statistical Analysis 1: Comparison: Fluticasone Furoate 110 mcg; Test type: Superiority or Other; p > 0.05, t-test, 2 sided — Comparison between Screening value and Visit 3 value

12. Primary Outcome: Creatinine Value at Baseline and After Treatment Completion
Description: Creatinine is a metabolic waste product in urine that remains relatively constant in an individual and that may be used to establish baseline renal function. Normal range: 53-100 umol/L (female) and 62-120 umol/L (male).
Time Frame: Baseline and treatment completion (up to Week 6)
Population: ITT Population
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Fluticasone Furoate 110 mcg
Number analyzed (Participants) | 56
umol/L
  Baseline | 90.21 (12.00)
  After treatment completion | 89.71 (15.21)
Statistical Analysis 1: Comparison: Fluticasone Furoate 110 mcg; Test type: Superiority or Other; p > 0.05, t-test, 2 sided — Comparison between Screening value and Visit 3 value

13. Primary Outcome: Alkaline Phosphatase Value at Baseline and After Treatment Completion
Description: Alkaline phosphatase is an enzyme produced by the liver or bone. An elevated level of alkaline phosphatase in the blood may indicate a liver or bone problem. Normal range: 30-120 units per liter (U/L).
Time Frame: Baseline and treatment completion (up to Week 6)
Population: ITT Population
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Fluticasone Furoate 110 mcg
Number analyzed (Participants) | 56
U/L
  Baseline | 73.05 (38.90)
  After treatment completion | 68.02 (18.53)
Statistical Analysis 1: Comparison: Fluticasone Furoate 110 mcg; Test type: Superiority or Other; p > 0.05, t-test, 2 sided — Comparison between Screening value and Visit 3 value

14. Primary Outcome: Aspartate Aminotransferase (AST) Value at Baseline and After Treatment Completion
Description: AST is a liver enzyme released into the blood when certain organs or tissues, particularly the liver and heart, are injured. Normal range: <=37 U/L.
Time Frame: Baseline and treatment completion (up to Week 6)
Population: ITT Population
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Fluticasone Furoate 110 mcg
Number analyzed (Participants) | 56
U/L
  Baseline | 26.50 (6.48)
  After treatment completion | 25.78 (4.18)
Statistical Analysis 1: Comparison: Fluticasone Furoate 110 mcg; Test type: Superiority or Other; p > 0.05, t-test, 2 sided — Comparison between Screening value and Visit 3 value

15. Primary Outcome: Alanine Aminotransferase (ALT) Value at Baseline and After Treatment Completion
Description: ALT is a liver enzyme that plays a role in protein metabolism. Abnormally high blood levels of ALT are a sign of liver inflammation or damage from infection or drugs. Normal range: <=40 U/L.
Time Frame: Baseline and treatment completion (up to Week 6)
Population: ITT Population
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Fluticasone Furoate 110 mcg
Number analyzed (Participants) | 56
U/L
  Baseline | 26.57 (16.36)
  After treatment completion | 24.29 (10.68)
Statistical Analysis 1: Comparison: Fluticasone Furoate 110 mcg; Test type: Superiority or Other; p > 0.05, t-test, 2 sided — Comparison between Screening value and Visit 3 value

16. Primary Outcome: Glucose Value at Baseline and After Treatment Completion
Description: Glucose is a simple sugar used as a source of energy for cellular metabolism. Normal range: 3.9-6.4 mmol/L.
Time Frame: Baseline and treatment completion (up to Week 6)
Population: ITT Population
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Fluticasone Furoate 110 mcg
Number analyzed (Participants) | 56
mmol/L
  Baseline | 5.07 (0.59)
  After treatment completion | 5.15 (0.53)
Statistical Analysis 1: Comparison: Fluticasone Furoate 110 mcg; Test type: Superiority or Other; p > 0.05, t-test, 2 sided — Comparison between Screening value and Visit 3 value

17. Primary Outcome: Urea Nitrogen Value at Baseline and After Treatment Completion
Description: The urea concentration of serum or plasma, conventionally specified in terms of nitrogen content and called blood urea nitrogen (BUN), is an important indicator of renal function. Normal range: 2.5-7.5 mmol/L.
Time Frame: Baseline and treatment completion (up to Week 6)
Population: ITT Population
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Fluticasone Furoate 110 mcg
Number analyzed (Participants) | 56
mmol/L
  Baseline | 5.78 (1.29)
  After treatment completion | 6.13 (1.40)
Statistical Analysis 1: Comparison: Fluticasone Furoate 110 mcg; Test type: Superiority or Other; p > 0.05, t-test, 2 sided — Comparison between Screening value and Visit 3 value

18. Primary Outcome: Total Protein Value at Baseline and After Treatment Completion
Description: A total protein assay measures the amount of proteins found in the plasma. Normal range: 65-82 g/L.
Time Frame: Baseline and treatment completion (up to Week 6)
Population: ITT Population
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Fluticasone Furoate 110 mcg
Number analyzed (Participants) | 56
g/L
  Baseline | 76.61 (4.15)
  After treatment completion | 76.89 (3.40)
Statistical Analysis 1: Comparison: Fluticasone Furoate 110 mcg; Test type: Superiority or Other; p > 0.05, t-test, 2 sided — Comparison between Screening value and Visit 3 value

19. Primary Outcome: Albumin Value at Baseline and After Treatment Completion
Description: Albumin is a simple water-soluble protein found in many tissues and liquids. Normal range: 35-50 g/L.
Time Frame: Baseline and treatment completion (up to Week 6)
Population: ITT Population
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Fluticasone Furoate 110 mcg
Number analyzed (Participants) | 56
g/L
  Baseline | 44.95 (2.04)
  After treatment completion | 45.22 (2.07)
Statistical Analysis 1: Comparison: Fluticasone Furoate 110 mcg; Test type: Superiority or Other; p > 0.05, t-test, 2 sided — Comparison between Screening value and Visit 3 value

20. Primary Outcome: Number of Participants With Normal and Abnormal Electrocardiogram (ECG) Results at Baseline and at Treatment Completion
Description: The electrocardiogram is a recording of the electrical activity of the heart as it undergoes excitation (depolarization) and recovery (polarization) to initiate each beat of the heart. Normal ECG readings show a slight flat-dip in between contractions and relaxations. An abnormal ECG is determined by comparing the results of an ECG graph with a standard or normal heart graph. If these flat-dips are not present, it may be an indication of a more serious problem.
Time Frame: Baseline and treatment completion (up to Week 6)
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Fluticasone Furoate 110 mcg
Number analyzed (Participants) | 56
participants
  Normal, Baseline | 56
  Abnormal, Baseline | 0
  Normal, At treatment completion | 56
  Abnormal, At treatment completion | 0

21. Primary Outcome: Percentage of Participants With Appearance of Nasal Polyps and Nasal Ulcers at Baseline and at Treatment Completion
Description: Nasal polyps are non cancerous growths occurring in the nose or sinuses. Nasal ulcers are a break in skin or mucous membrane with loss of surface tissue, disintegration and necrosis of epithelial tissue.
Time Frame: Baseline and treatment completion (up to Week 6)
Population: ITT Population
Measure: Number; unit: percentage of participants
Arm/Group | Fluticasone Furoate 110 mcg
Number analyzed (Participants) | 56
percentage of participants
  Baseline, nasal polyps | 0
  After treatment completion, nasal polyps | 0
  Baseline, nasal ulcers | 0
  After treatment completion, nasal ulcers | 0

ADVERSE EVENTS:
Time Frame: During treatment period and a phone call questioning participants about adverse events 3-5 days after the end of study treatment (up to week 7)
Description: Serious adverse events (SAEs) and adverse events (AEs) were collected in the ITT Population.
Arm/Group | Fluticasone Furoate 110 mcg
Serious Adverse Events (participants affected / at risk) | 0/56
Other Adverse Events (participants affected / at risk) | 13/56
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fluticasone Furoate 110 mcg (N=56)
Headache (General disorders) | 1
Migraine (Nervous system disorders) | 1
Menorrhagia (Reproductive system and breast disorders) | 1
Fatigue (General disorders) | 1
Sleepy (General disorders) | 1
Ear pain (Ear and labyrinth disorders) | 1
Dry nose (Respiratory, thoracic and mediastinal disorders) | 1
Burning urination (Renal and urinary disorders) | 1
Eyelid swelling (Eye disorders) | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1
Itchy nose (Respiratory, thoracic and mediastinal disorders) | 1
Sneeze (Respiratory, thoracic and mediastinal disorders) | 1
Congested nose (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.